CLINICAL TRIAL: NCT07226674
Title: MAEVE: Microbiota Mediated Flavonoid Metabolites for Cognitive Health
Brief Title: Microbiota Mediated Flavonoid Metabolites for Cognitive Health
Acronym: MAEVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: University of Parma (Other); University College Cork (Other); National Institute on Aging (NIA) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/25/0046; 1R01AG081768-01 (NIH); 5R01AG081768-02 (NIH)
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Decline; Cognitive Dysfunction
Keywords: Polyphenols; Mediterranean Diet; Gut Microbiome; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Interventional Model
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenol Supplement (Experimental): Juice Plus Essentials, Berry Blend Capsules
  Interventions: Dietary Supplement: Polyphenol Supplement
- Placebo Supplement (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Polyphenol Supplement — Juice Plus Essentials, Berry Blend Capsules
  Arms: Polyphenol Supplement
Dietary Supplement: Placebo Supplement — Micronutrient matched placebo
  Arms: Placebo Supplement

SUMMARY:
Globally, populations are ageing increasing the prevalence of Alzheimer's disease (AD), due to lack of effective treatments. The traditional Mediterranean diet, rich in fibre and polyphenols (PPs) can help prevent or delay cognitive dysfunction and preserve healthy brain structure and function. Cognitive decline is inversely associated with higher PP intakes (>421mg/day) i.e., total flavonoids, flavan-3-ols and flavonoid oligomers. The positive brain effects of flavonoid intake are likely mediated in part by gut microbial PP metabolites, consistent with the emerging role of the brain-gut microbiome (BGM) system in neurodegeneration. Our preliminary data indicate that circulating phenyl-γ-valerolactones (PVL), neuroprotective compounds exclusively produced by gut microbiota from flavan-3-ol rich foods18 are associated with delaying cognitive dysfunction. Intake of PPs change gut microbial composition and function, altering the physiology of the host's secondary bile acid (BA) pool through modulation of bacterial 7α-dehydroxylation of de-conjugated primary BAs into secondary BAs. This is noteworthy as 7α-dehydroxylation of BAs does not happen in the brain and because gut microbial BA metabolites have regulatory and signalling functions in the brain. The ratio between certain primary and secondary BAs is also dysregulated in AD with significantly lower serum concentrations of cholic acid (a primary BA) and increased levels of deoxycholic acid (a bacterially produced secondary BA). The increased ratio of cholic acid to deoxycholic acid is correlated with cognitive decline. Increased levels of tyrosine, tryptophan, purine, and tocopherol have also been identified in postmortem AD brains. However, specific pathways and mechanisms underlying these associations are unclear. In this multi-PI application by leaders in the field of BGM interactions, we leverage the collectively (NIH, HSC, SFI) funded Tripartite US-Ireland R&D Partnership Program to determine the mechanisms involved in PP intake on maintaining healthier cognitive and brain function, as mediated by gut microbiota metabolites of PP and BAs in 50+ year old elderly with enhanced AD risk.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years
* BMI ≥ 25 kg/m2
* Enhanced risk of AD - defined as family history of AD, 1st degree family member
* Habitually consume suboptimal diets such as typical Western diet (i.e., high in animal products, refined carbohydrates and processed food).
* Subjects capable of and willing to comply with the protocol and to give their written informed consent.

Exclusion Criteria:

* Cognitive impairment at time of recruitment into the study, as measured by the Mini Mental Status Exam (MMSE, score 25-30), and Clinical Dementia Rating (CDR, score=0) or Everyday Cognition Scale-12 (ECog-12, score<1.36 included).
* Pre-existing psychosis or psychiatric conditions.
* Currently receiving treatment for dementia.
* History of substance abuse or cerebrovascular events.
* Heavy use of tobacco (>1/2 pack per day)
* Any intolerance or allergy documented or suspected to one of the components of the study products.
* Have taken probiotics or antibiotic therapy within the last 1 month
* Change in medication use in the last 3 months.
* Frailty, malnutrition, or food allergy/intolerance requiring special diets will also be excluded.
* Following any specific diet (vegetarian, vegan, etc.)
* Body weight at enrolment greater than 400lbs due to weight restrictions on the MRI table.
* Pregnant, breastfeeding, postpartum for less than 6 months, or unwilling to practice birth control during participation in the study.
* Unable to safely participate in the MRI (claustrophobia, presence of devices affected by MRI such as pacemakers, neurostimulators, or metallic foreign body, etc.)
* Chronic pain.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Having a psychological or linguistic inability to sign the informed consent;
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Subject participating in another biomedical study or participation in another study within the 3 months before entry into this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Differences in Polyphenol-derived metabolite concentrations pre, mid, & post intervention - stool | Collected three times by the participant at home, once at baseline (week 0), once at mid-study (month 6), and once at the final 12month appointment (month 12)
  Measurement of metabolomics via stool specimen.
Differences in Polyphenol-derived metabolite concentrations pre, mid, & post intervention - blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of metabolomics via blood specimen.
Differences in microbiome levels pre, mid, & post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  16S RNA sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  16S RNA sequencing to measure microbiome levels via blood specimen.
Differences in microbiome levels pre, mid, & post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via stool specimen.
Differences in microbiome levels pre, mid, & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Shotgun metagenomics, sequencing to measure microbiome levels via stool specimen.
Differences in Cognitive Measures pre, mid, & post intervention - Executive Function | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized Stroop Neuro-psychological test; participants ability to correctly identify colours when words are printed in conflicting ink colours.
Differences in Cognitive Measures pre, mid, & post intervention - Executive Function | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized Trails A & B; participants ability to connect dots, in order, as quickly as possible.
Differences in Cognitive Measures pre, mid, & post intervention | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Differences in Cognitive Measures pre, mid, & post intervention | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Administration of a standardized arithmetic task; participants ability to complete quick mental math.

SECONDARY OUTCOMES:
Differences in tryptophan-associated metabolite profiles pre, mid, and post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of tryptophan-associate metabolite profiles via stool specimen.
Differences in Bile Acid's (BA's) pre, mid, & post intervention - Stool | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of BA's via stool specimen.
Differences in Inflammatory markers pre, mid, & post intervention - Blood | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of inflammatory markers via blood specimen.
Differences in Alzheimer's Disease (AD) markers pre, mid, & post intervention - Blood [Time | Collected three times, once at baseline appointment (week 0), once at mid-study appointment (month 6), and once at the final 12month appointment (month 12).
  Measurement of AD markers via blood specimen.
Anthropometrics - BMI | Measured three times, once at each in-clinic appointment (week 0, month 6, month 12)
  Measurement of height(in) and weight(lbs), used to calculate body mass index (BMI)
Questionnaire Data | Collected 3 times (1) before beginning the dietary supplement, (2) mid-study month 6, (3) end of study month 12.
  Use of validated surveys to assess ingestive behaviours, social isolation, stress, health, physical activity, etc., self-reported by the participant at home.
Monthly Questionnaire Data | Collected 3 times (1) before beginning the dietary supplement, (2) mid-study month 6, (3) end of study month 12.
  Collected once a month for the duration of the study (12months).
Anthropometrics - waist and hip circumference | Measured three times, once at each in-clinic appointment (week 0, month 6, & month 12)
  Measurement of waist and hip circumference (cm)
Systolic and Diastolic Blood Pressure | Measured three times, once at each in-clinic appointment (week 0, month 6, month 12).
  Measurement of the pressure of circulating blood at rest

OTHER OUTCOMES:
Differences in Multimodal Brain Signatures pre, mid, & post intervention | Measured thrice, once at baseline (week 0), mid-study (month 6), and final 12month appointment (month 12) visit.
  Neuroimaging of participants brain via magnetic resonance imaging (MRI) procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gill, PhD, Principal Investigator — Ulster University, Human Intervention Studies Unit, Coleraine, Co. Londonderry, BT52 1SA, United Kingdom.
Locations (1):
- Ulster University, Human Intervention Studies Unit, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No